CLINICAL TRIAL: NCT03851133
Title: The Florida Pancreas Collaborative Next-Generation Biobank: Reducing Health Disparities and Improving Survival for Pancreatic Cancer
Brief Title: Florida Pancreas Collaborative Next Generation Biobank
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-19717; 8JK02 (Other: Florida Department of Health)
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Cancer Cachexia
Keywords: pancreas; biobank; quantitative imaging; biomarkers; health disparities
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Serum, Tumor tissue from biopsy or surgery, Muscle and fat tissue from surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Blood samples, tumor samples and data will be collected from all participants as applicable.
  Interventions: Other: Blood Sample Collection; Other: Tumor Sample collection; Other: Data Collection

INTERVENTIONS:
Other: Blood Sample Collection — Participants will be asked to donate blood at baseline (+/- 30 days of diagnosis date) and at the time of follow-up (approximately 6 months and approximately 12 months after baseline).
Other: Tumor Sample collection — At the time of tissue biopsy and surgical resection (if applicable), pancreatic tumor tissue and tissue from site of metastasis will be collected.
Other: Data Collection — Participants will be asked to complete a 3 page screening tool at the time of their in-person clinic visit, as well as questionnaires at baseline and at 6 and 12 months.

SUMMARY:
The goal of this study is to partner with individuals known or suspected to have pancreatic cancer to build a biobank dedicated to minimizing disparities and personalizing care for individuals affected by pancreatic cancer. A biobank is a resource that involves collection, processing and storage of blood, other bodily fluids, and tissue.

DETAILED DESCRIPTION:
Doctors, researchers, and patient advocates from numerous institutions throughout the state of Florida have formed a partnership known as the Florida Pancreas Collaborative. The goals of the Florida Pancreas Collaborative team are to find better ways to diagnose and treat pancreatic cancer and improve quality of life. Recent research suggests that pancreatic cancer affects people of various racial and ethnic groups differently, with some groups having more aggressive disease and a poorer prognosis than other groups.

In this research study, the investigators want to partner with individuals known or suspected to have pancreatic cancer to build a 'biobank' dedicated to minimizing disparities and personalizing care for individuals affected by pancreatic cancer. A biobank is a valuable resource that involves collection, processing, and storage of blood, other bodily fluids, and tissue (obtained during biopsy or surgery) to improve the investigator's understanding of health and disease. When combined with information and medical images obtained through routine care, the investigators will be able to investigate biological processes that may underlie differences and poor outcomes and target them with more effective therapeutic strategies tailored to the individual.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Patient presents for evaluation at a participating site with a strong clinical suspicion or diagnosis of a pancreatic cancer primary based on symptoms, imaging, biopsy, and/or blood-work and has not had treatment.
* Patient self-reports as Non-Hispanic White, African American, or Hispanic.
* Able to understand and voluntarily sign the informed consent.
* Willing to complete study questionnaire(s) and donate medical images and biological specimens (including tissue and blood) obtained at the time of standard of care procedures (biopsy, surgery, and/or venipuncture) after signing the informed consent document.

Exclusion Criteria:

* No suspicion or diagnosis of pancreatic cancer.
* Has a diagnosis of pancreatic cancer but and has already undergone treatment (which may include surgery, chemotherapy, and/or radiation).
* Self-reported race/ethnicity other than Non-Hispanic White, African American, or Hispanic.
* Unable to provide informed consent.
* Unwilling to complete study questionnaires(s) and/or donate biological specimens

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting at any of the participating sites with a diagnosis or suspicion or pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of Precachexia | Up to 12 months
  Cases will be evaluated for precachexia using the following guidelines: Anorexia with <5% weight loss over past 6 months along with metabolic changes that together indicate precachexia.
Evidence of Cachexia | Up to 12 months
  Cases will be evaluated for cachexia using the following guidelines: Anorexia with >5% weight loss over past 6 months, along with metabolic changes that together indicate cachexia.
Evidence of Refractory Cachexia | Up to 12 months
  Cases will be evaluated for refractory cachexia using the following guidelines: Anorexia >5% weight loss over 6 months along with specific metabolic changes that together indicate refractory cachexia.
Presence of Myopenia | Up to 12 months
  Measures of skeletal muscle index (SMI) and psoas muscle index (PMI) for will be used for myopenia assessment.
Presence of Visceral Adiposity | Up to 12 months
  Using CT scans at the axial L2-L3 level, the following radiologic measures of abdominal adiposity will be obtained: visceral fat area (VFA), subcutaneous fat area (SFA), total abdominal fat (TAF) area, and the VFA to SFA ratio (V/S). The VFA to SFA ratio (V/S) will be calculated with V/S > 0.4 defined as viscerally obese.

SECONDARY OUTCOMES:
Overall Survival | Up to 24 months
  Overall Survival will be defined as time from surgery to death from any cause
Progression Free Survival | Up to 24 months
  Progression Free Survival will be defined as time from surgery to pancreatic cancer recurrence or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Permuth, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (14):
- United States (14):
  - Lee Memorial Hospital Regional Cancer Center, Fort Myers, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Palmetto General Hospital, Hialeah, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Lakeland Regional Health, Lakeland, Florida
  - Sylvester Comprehensive Cancer Center & Jackson Memorial Hospital, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Advent Health - Orlando, Orlando, Florida
  - University of Florida - Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St Anthony's Baycare/Bay Surgical Specialists, St. Petersburg, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - University of South Florida/Tampa General Hospital, Tampa, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
Investigators requesting to use Florida Pancreas Collaborative (FPC) data, images, and/or biospecimens will need to submit a written proposal to the FPC biobank utilization committee. Decisions will be based on scientific merit, specimen availability, experience of the requesting investigator, and resources to conduct proposed methods. De-identified samples and/or data will be released if the concept receives approval and after scientific review committee and IRB approval is obtained, conflict of interests are checked, and a material transfer agreement is established. Intellectual property issues will need to be agreed upon. If access is granted, the biobank utilization committee may monitor the Investigator's Research studies to ensure appropriate use of the biospecimens and/or data. The Investigator shall provide a written summary of their research findings and reference this funding source in future manuscripts and presentations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be available approximately one year after study ends, approximately September 2022. End of availability undetermined at this time.
Access Criteria: Data and specimens will be shared with researchers interested in this topic area who wish to pursue analyses that may be descriptive, analytic, molecular, or correlative in nature. The access criteria used to share IPD and any additional supporting information will involve a formal process which involves submitting a written proposal to the FPC biobank utilization committee. Decisions will be based on scientific merit, specimen availability, experience of the requesting investigator, and resources to conduct proposed methods. Samples and/or data will be released if the concept receives approval and after scientific review committee and IRB approval is obtained, conflict of interests (COI) are checked, a material transfer agreement is established between institutions, and intellectual property issues are agreed upon. The release of data will be based on the nature of the request and can represent aggregate or individual-level data.